CLINICAL TRIAL: NCT07353229
Title: Phase 1 Trial of 68Ga-Dotatate PET and MRI Guided Radiation Dose Escalation for High-Risk Meningiomas
Brief Title: 68Ga-Dotatate PET and MRI Guided Radiation Dose Escalation for High Risk Meningioma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: dose escalation trial, and the first 3 patients (who made up a cohort) were all accrued
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: iRIS ID-2023-2983; JT 38404 (Other: JeffTrial Number)
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: High Risk Meningioma; Recurrent Meningioma
Keywords: High-Risk Meningiomas; subtotal resection of Grade 2 meningioma; subtotal resection of Grade 3 meningioma; recurrent meningioma; 68Ga-Dotatate PET; MRI Guided Radiation; BOIN; maximum tolerated dose
MeSH Terms: conditions — Meningioma | interventions — Magnetic Resonance Imaging; Surveys and Questionnaires; Fertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1: Dose Level 1 - 66 Gy (Experimental): Participants receive 68Ga-Dotatate PET and MRI guided external beam radiation therapy (EBRT) with intensity-modular radiation therapy (IMRT) or volumetric arc radiation therapy (VMAT). Two planning target volumes (PTV) will be required, including PTV and PTV-high. PTV_High will be given a dose of 66 Gy in 30 once daily fractions. PTV will receive 60 Gy in 30 fractions concurrently.
  Interventions: Radiation: ⁶⁸Ga-Dotatate PET and MRI Guided Radiation Therapy; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: 68Ga-Dotatate PET Imaging; Other: MD Anderson Symptom Inventory Bain Tumor form (MDASI-BT); Diagnostic Test: EuroQol-5 Dimension (ED-5D)
- Arm 2: Dose Level 2 - 69 Gy (Experimental): Participants receive 68Ga-Dotatate PET and MRI guided external beam radiation therapy (EBRT) with intensity-modular radiation therapy (IMRT) or volumetric arc radiation therapy (VMAT). Two planning target volumes (PTV) will be required, including PTV and PTV-high. PTV_High will be given a dose of 69 Gy in 30 once daily fractions. PTV will receive 60 Gy in 30 fractions concurrently.
  Interventions: Radiation: ⁶⁸Ga-Dotatate PET and MRI Guided Radiation Therapy; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: 68Ga-Dotatate PET Imaging; Other: MD Anderson Symptom Inventory Bain Tumor form (MDASI-BT); Diagnostic Test: EuroQol-5 Dimension (ED-5D)
- Arm 3: Dose Level 3 - 72 Gy (Experimental): Participants receive 68Ga-Dotatate PET and MRI guided external beam radiation therapy (EBRT) with intensity-modular radiation therapy (IMRT) or volumetric arc radiation therapy (VMAT). Two planning target volumes (PTV) will be required, including PTV and PTV-high. PTV_High will be given a dose of 72 Gy in 30 once daily fractions. PTV will receive 60 Gy in 30 fractions concurrently.
  Interventions: Radiation: ⁶⁸Ga-Dotatate PET and MRI Guided Radiation Therapy; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: 68Ga-Dotatate PET Imaging; Other: MD Anderson Symptom Inventory Bain Tumor form (MDASI-BT); Diagnostic Test: EuroQol-5 Dimension (ED-5D)
- Arm 4: Dose Level 4 - 75 Gy (Experimental): Participants receive 68Ga-Dotatate PET and MRI guided external beam radiation therapy (EBRT) with intensity-modular radiation therapy (IMRT) or volumetric arc radiation therapy (VMAT). Two planning target volumes (PTV) will be required, including PTV and PTV-high. PTV_High will be given a dose of 75 Gy in 30 once daily fractions. PTV will receive 60 Gy in 30 fractions concurrently.
  Interventions: Radiation: ⁶⁸Ga-Dotatate PET and MRI Guided Radiation Therapy; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: 68Ga-Dotatate PET Imaging; Other: MD Anderson Symptom Inventory Bain Tumor form (MDASI-BT); Diagnostic Test: EuroQol-5 Dimension (ED-5D)
- MTD Expansion Cohort (Experimental): Once the maximum tolerated dose (MTD) is established, an additional 12 patients will be enrolled at that dose level. Participants will receive 68Ga-Dotatate PET imaging and MRI-guided external beam radiation therapy (EBRT), delivered using either intensity-modulated radiation therapy (IMRT) or volumetric modulated arc therapy (VMAT). Two planning target volumes (PTVs) will be defined: PTV and PTV-High. PTV-High will receive the MTD (in Gy) delivered in 30 once-daily fractions. PTV will concurrently receive 60 Gy in 30 fractions.
  Interventions: Radiation: ⁶⁸Ga-Dotatate PET and MRI Guided Radiation Therapy; Diagnostic Test: Magnetic Resonance Imaging (MRI); Diagnostic Test: 68Ga-Dotatate PET Imaging; Other: MD Anderson Symptom Inventory Bain Tumor form (MDASI-BT); Diagnostic Test: EuroQol-5 Dimension (ED-5D)

INTERVENTIONS:
Radiation: ⁶⁸Ga-Dotatate PET and MRI Guided Radiation Therapy — The radiation dose levels will be 66, 69, 72, and 75 Gy in 30 daily fractions based on the design.
Diagnostic Test: Magnetic Resonance Imaging (MRI) — MRI brain with and without contrast must be performed within 6 weeks prior to registration. MRI brain will be performed at 3-, 6-, 9-, 12-, 18-, and 24 months. If surgery is performed, MRI must be performed after surgery.
  Other Names: MRI
Diagnostic Test: 68Ga-Dotatate PET Imaging — ⁶⁸(GA)Dotatate PET must be performed within 6 weeks prior to registration. 12 months after radiation treatment +/- 1 month patients are required to get Ga-Dotatate PET.
  Other Names: GaTate PET; Gallium-68 DOTATATE Scan; DOTA-TATE imaging
Other: MD Anderson Symptom Inventory Bain Tumor form (MDASI-BT) — Every 3 m ± 2 weeks, starting 3 m ± 2 weeks post radiation treatment. MRI at the 9 month post radiation visit is only to be completed if per physician discretion it is clinically indicated, except for patients with grade 3 meningioma, the 9 month MRI is required. At month 18 ± 4 weeks, and month 24 ± 4 weeks after radiation treatment.
  Other Names: Survey
Diagnostic Test: EuroQol-5 Dimension (ED-5D) — Every 3 m ± 2 weeks, starting 3 m ± 2 weeks post radiation treatment. MRI at the 9 month post radiation visit is only to be completed if per physician discretion it is clinically indicated, except for patients with grade 3 meningioma, the 9 month MRI is required. At month 18 ± 4 weeks, and month 24 ± 4 weeks after radiation treatment.
  Other Names: Survey

SUMMARY:
The is phase 1 trial of 68Ga-Dotatate PET/MRI guided radiation dose escalation for high-risk meningiomas (defined as recurrent or subtotal resection of Grade 2, and any Grade 3 meningioma). A modified toxicity probability interval schedule will be implemented with a Bayesian Optimal interval suite. It includes 4 dose cohort (66 Gy, 69 Gy, 72 Gy and 75 Gy). The initial study cohort will include 3 patients treated with 69 Gy in 30 daily fractions. The investigators will seek to determine the MTD of radiation therapy based DLTs.

DETAILED DESCRIPTION:
Patient will be enrolled, and dose selected per modified toxicity probability interval utilizing a Bayesian Optimal interval suite to maximize the probability that selecting the MTD dose that has a target DLT rate under 30% while optimizing patient safety over the 3+3 trial design 15. For our initial cohort the investigators will seek to treat 3 patients at 69 Gy in 30 daily fractions, Monday-Friday for 6 weeks of treatment utilizing MRI/PET target delineation with IMRT/VMAT. Patients will be followed weekly for on-treatment visits and 30 days from end of radiation to evaluate for DLTs classified as grade 3+ toxicity by NCI-CTCAE v5.0. Subsequent dosing will be determined by DLTs experienced utilizing a modified toxicity probability interval design. If the stopping rule is met, the trial will discontinue enrollment and select the MTD. If the stopping rule is not met, the DLT rate will be computed at the current treated dose. DLT rate is calculated by the total number of patients experiencing DLT at the current dose divided by total number of evaluable patients at the current dose. With a DLT rate of less than or equal to 0.236 dose will be escalated by 3 Gy, DLT rate greater than 0.359 will de-escalate the dose by 3 Gy. A rate between 0.236 and 0.359 will retain the current dose. An additional 3 patients will then be enrolled at specified dose depending on DLT rate. Patients will be treated and followed to assess for acute DLTs. The process will be repeated with enrollment discontinued if stopping rule met or additional patient will be enrolled at a dose from 66 - 75 Gy in 30 fractions based on new DLT rate. Enrollment utilizing DLT rate will be discontinued once stopping rule met or 12 patients are enrolled and an MTD will be established. Once the MTD has been established, an additional 12 patients at the MTD will then be enrolled.

Following radiation treatment (with once weekly on-treatment visits) and evaluation 1 month following completion for radiation, patients will be evaluated 3-, 6-, 9, 12-, 18-, and 24-months post-treatment utilizing NCI-CTCAEv5.0, symptom burden and QOL questionnaires, and MRI imaging to evaluate for safety, toxicity, and treatment efficacy.

The study population will include any adult patients, with high-risk meningioma as defined by RTOG definition (Grade 2 meningioma with subtotal resection or recurrence, and any Grade 3 meningioma).

It is believed dose escalation with IMRT/VMAT therapy is feasible and well tolerated with improved target delineation utilizing both MRI and PET fusion with an acceptable toxicity profile.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all the following inclusion criteria in order to be eligible to participate in the study:

  1. Adult patients, age ≥ 18 years
  2. Patients with RTOG Group III meningioma (high risk) defined as:

     * Patients with newly diagnosed or a recurrent WHO grade 3 meningioma of any resection extent.
     * or patients with a recurrent WHO grade 2 meningioma of any resection extent.
     * or patient with a newly diagnosed sub-totally resected (residual nodular enhancement or PET enhancement on postoperative imaging, or Simpson grade IV or V excision) WHO grade 2 meningioma.
  3. In the setting of newly diagnosed meningioma, the histologic diagnosis must be within 6 months of registration.
  4. In the setting of a recurrent meningioma, there are no such time constraints. However, additional resection or biopsy is encouraged for patients with recurrence but is not requisite. If further biopsy or resection is performed at recurrence, it must be within 6 months of registration.
  5. Karnofsky Performance Status 60-100
  6. MRI brain and ⁶⁸Ga-Dotatate PET must be performed within 6 weeks prior to registration.
  7. For woman of childbearing potential:

     * A negative serum pregnancy test is required within 14 days prior to registration.
     * The patient must agree to practice adequate contraception from the time of the negative serum pregnancy test throughout the entire course of EBRT.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. Extracranial meningioma
  2. Prior radiation therapy to the scalp, cranium, brain, or skull base
  3. Prior malignancy (except for non-melanomatous skin cancer), unless disease free for at least 3 years
  4. Pregnancy or lactation
  5. Treatment with another investigational drug or other intervention at time of registration
  6. Inability to receive gadolinium or undergo MRI brain or ⁶⁸Ga-Dotatate PET imaging.
  7. Serious medical or psychiatric illness likely to interfere with participation in this clinical trial.
  8. Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema)
  9. Uncontrolled seizure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of 68Ga-Dotatate PET/MRI guided radiation dose escalation | 30 days post-treatment
  To establish MTD utilizing DLT rates (DLT will be defined as radiation treatment related G3 or higher neurological toxicity from beginning of radiation till 30 days after finishing radiation treatment).

SECONDARY OUTCOMES:
Late Neurological Toxicities of Radiation Treatment | up to 2 year post-treatment
  Number of participants experiencing radiation treatment related G3 or higher neurological toxicity from beginning of radiation till 30 days after finishing radiation treatment.
Symptom Burden Assessment Using MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire | Baseline
  Patient reported symptom severity and interference will be assessed using the MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire. It consists of 23 symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours. The interference items also are measured on 0-10 scales.
Symptom Burden Assessment Using MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire | 3 months (+/- 2 weeks)
  Patient reported symptom severity and interference will be assessed using the MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire. It consists of 23 symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours. The interference items also are measured on 0-10 scales.
Symptom Burden Assessment Using MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire | 6 months (+/- 2 weeks)
  Patient reported symptom severity and interference will be assessed using the MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire. It consists of 23 symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours. The interference items also are measured on 0-10 scales.
Symptom Burden Assessment Using MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire | 9 months (+/- 2 weeks)
  Patient reported symptom severity and interference will be assessed using the MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire. It consists of 23 symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours. The interference items also are measured on 0-10 scales.
Symptom Burden Assessment Using MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire | 12 months (+/- 2 weeks)
  Patient reported symptom severity and interference will be assessed using the MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire. It consists of 23 symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours. The interference items also are measured on 0-10 scales.
Symptom Burden Assessment Using MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire | 18 months (+/- 4 weeks)
  Patient reported symptom severity and interference will be assessed using the MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire. It consists of 23 symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours. The interference items also are measured on 0-10 scales.
Symptom Burden Assessment Using MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire | 24 months (+/- 4 weeks)
  Patient reported symptom severity and interference will be assessed using the MD Anderson Symptom Inventory - Brain Tumor (MDASI - BT) Questionnaire. It consists of 23 symptoms rated on an 11-point scale (0 to 10) to indicate the presence and severity of the symptom, with 0 being "not present" and 10 being "as bad as you can imagine." Each symptom is rated at its worst in the last 24 hours. The interference items also are measured on 0-10 scales.

OTHER OUTCOMES:
Local Control at 1 year from Registration | at 1 year from Registration
  Proportion of participants without local tumor progression.
Local Control at 2 years from Registration | at 2 years from Registration
  Proportion of participants without local tumor progression.
Local Control at 3 years from Registration | at 3 years from Registration
  Proportion of participants without local tumor progression.
Progression Free Survival at 1 year from Registration | at 1 year from Registration
  Time from enrollment to disease progression or death from any cause, whichever occurs first.
Progression Free Survival at 2 years from Registration | at 2 years from Registration
  Time from enrollment to disease progression or death from any cause, whichever occurs first.
Progression Free Survival at 3 years from Registration | at 3 years from Registration
  Time from enrollment to disease progression or death from any cause, whichever occurs first.
Overall Survival at 1 year from Registration | at 1 year from Registration
  Time from enrollment to death from any cause.
Overall Survival at 2 years from Registration | at 2 years from Registration
  Time from enrollment to death from any cause.
Overall Survival at 3 years from Registration | at 3 years from Registration
  Time from enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, PhD, Principal Investigator — Wenyin.Shi@jefferson.edu
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States